CLINICAL TRIAL: NCT02500082
Title: Compassionate Use of Triheptanoin (UX007) to Treat Citrate Transporter Deficiency
Brief Title: Triheptanoin (UX007) to Treat Citrate Transporter Deficiency
Status: No longer available | Type: Expanded Access
Sponsor: Irina A Anselm (Other)
Responsible Party: Sponsor-Investigator, Irina A Anselm, Assistant in Neurology, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Other Study IDs: IRB-P00017250
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Citrate Transporter Deficiency; SLC13A5 Gene Mutation
Keywords: citrate transporter deficiency; SLC13A5 gene; citric acid cycle; energy metabolism
MeSH Terms: interventions — triheptanoin

INTERVENTIONS:
Drug: triheptanoin — Triheptanoin (UX007) is a medium chain triglyceride of three seven-carbon fatty acids (C7), on a glycerol backbone, with a molecular formula of C24H44O6. It is being evaluated as a substrate replacement therapy for the treatment of long-chain fatty acid oxidation disorders (LC-FAOD) and for the treatment of seizures associated with Glut 1 DS. Triheptanoin is metabolized to provide substrate replacement for both fatty acid metabolism and anaplerosis (replacement of TCA cycle intermediates) required to restore the efficient generation of energy and the net production of glucose in patients. The mechanism of action of triheptanoin in restoring energy metabolism is dependent on its medium-chain length as well as its odd-carbon properties. Triheptanoin is a highly purified form intended for oral administration.
  Other Names: UX007

SUMMARY:
The purpose of this study is to determine whether triheptanoin (UX007) is effective in the treatment of neurological symptoms related to citrate transporter deficiency (SLC13A5 gene mutation).

DETAILED DESCRIPTION:
This compassionate use research study has been developed to study an investigational drug, triheptanoin (UX007), for the treatment of neurological symptoms related to citrate transporter deficiency, a disease with no existing treatment. The hypothesis is that triheptanoin will restore deficient energy metabolism in these patients, leading to improved seizure control, mental clarity, and physical strength.

Based on the literature, the SLC13A5 gene product is a citrate transporter. However, there is the possibility that other compounds are transported as well. The gene may be expressed in human neurons and function at the level of the plasma membrane. The hypothesis is that the transport of citrate across the plasma membrane from the extracellular space into the cytoplasm plays a role in maintaining the pool size of citrate in both the cytoplasm and mitochondrial matrix. Triheptanoin therapy may increase the metabolism of odd-chain fatty acids in neuronal mitochondria and thereby increase the levels of succinyl-CoA, leading to an increase in citrate concentrations. The increased level of citrate in the mitochondrial matrix may lead to an increased efflux of citrate from the matrix to the cytoplasm, thus increasing the cytoplasmic pool of citrate and allowing the malfunctioning citrate transporter to be bypassed. If successful, triheptanoin treatment will improve neuronal function and lead to an improvement in CNS function for patients.

While investigators will follow the course of subjects with considerable interest and may use some of the collected data for clinical research, this study is done for humanitarian reasons.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of citrate transporter deficiency due to mutations in the SLC13A5 gene.
* Presentation with severe global developmental delay and seizures.

Exclusion Criteria:

* Valproate is an AED that partially inhibits the TCA cycle via alpha-ketoglutarate dehydrogenase and should not be administered to subjects taking UX007.

Ages: 4 Years to 9 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Irina A Anselm, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Department of Neurology, Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Johannessen CU, Petersen D, Fonnum F, Hassel B. The acute effect of valproate on cerebral energy metabolism in mice. Epilepsy Res. 2001 Dec;47(3):247-56. doi: 10.1016/s0920-1211(01)00308-4. PMID 11738932
- [Background] Pascual JM, Liu P, Mao D, Kelly DI, Hernandez A, Sheng M, Good LB, Ma Q, Marin-Valencia I, Zhang X, Park JY, Hynan LS, Stavinoha P, Roe CR, Lu H. Triheptanoin for glucose transporter type I deficiency (G1D): modulation of human ictogenesis, cerebral metabolic rate, and cognitive indices by a food supplement. JAMA Neurol. 2014 Oct;71(10):1255-65. doi: 10.1001/jamaneurol.2014.1584. PMID 25110966
- [Background] Thevenon J, Milh M, Feillet F, St-Onge J, Duffourd Y, Juge C, Roubertie A, Heron D, Mignot C, Raffo E, Isidor B, Wahlen S, Sanlaville D, Villeneuve N, Darmency-Stamboul V, Toutain A, Lefebvre M, Chouchane M, Huet F, Lafon A, de Saint Martin A, Lesca G, El Chehadeh S, Thauvin-Robinet C, Masurel-Paulet A, Odent S, Villard L, Philippe C, Faivre L, Riviere JB. Mutations in SLC13A5 cause autosomal-recessive epileptic encephalopathy with seizure onset in the first days of life. Am J Hum Genet. 2014 Jul 3;95(1):113-20. doi: 10.1016/j.ajhg.2014.06.006. PMID 24995870